CLINICAL TRIAL: NCT03007927
Title: Evaluation of Dexamethasone Added to the Usual Infiltration With Bupivacaine in Inguinal Hernia Repair Mesh
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SEBASTIAN ROCHE (Other)
Collaborators: Sebastián Roche, MD (Unknown); Santiago Bertone, MD (Unknown); Claudio Brandi, MD (Unknown)
Responsible Party: Sponsor-Investigator, SEBASTIAN ROCHE, Medical Doctor, Hospital Italiano de Buenos Aires
Organization: Hospital Italiano de Buenos Aires (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2736
Record Dates: First submitted 2016-12-20; First posted 2017-01-02 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2017-08

CONDITIONS: Pain, Postoperative
Keywords: pain; hernia repair; Dexamethasone
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine-Dexamethasone (Experimental): bupivacaine 1,5 mg/kg + dexamethasone 8 mg 2ml
  Interventions: Drug: Bupivacaine-Dexamethasone
- Bupivacaine- physiological solution (Active Comparator): bupivacaine 1,5 mg/kg + physiological solution
  Interventions: Drug: Bupivacaine- physiological solution

INTERVENTIONS:
Drug: Bupivacaine-Dexamethasone — Bupivacaine 1,5 mg/kg-Dexamethasone 2ml 8 mg
  Arms: Bupivacaine-Dexamethasone
Drug: Bupivacaine- physiological solution — Bupivacaine 1,5 mg/kg- physiological solution
  Arms: Bupivacaine- physiological solution

SUMMARY:
To evaluate the impact on the postoperative pain of the dexamethasone addition to the usual treatment with bupivacaine in the local infiltration of the surgical area in Inguinal Hernia Repair Mesh

DETAILED DESCRIPTION:
This study will be: controlled, prospective, randomized and double blind.

Randomized experimental study in which all patients scheduled to undergo unilateral inguinal hernia repair and who meet the inclusion criteria and none of the exclusion criteria will be invited to participate. At the time of admission to the study, they were assigned randomly to one of the two branches of intervention:

(Group A): infiltration with 0.5% bupivacaine in doses of 1.5 mg / kg body weight diluted in physiological solution to a final volume of 30 ml.

(Group B): infiltration with 0.5% bupivacaine at doses of 1.5 mg / kg body weight + dexamethasone 2 ml (8 mg) diluted in physiological solution to a final volume of 30 ml.

Pain will be evaluated through the visual analogue scale of 0-10 measured at the 1st postoperative hour, then every 2 hours until discharge, at discharge, at 8 hours, at 24 hours, 48 hours and at 8 days .

It will also evaluate analgesic consumption, complications and labor return

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years.
2. Unilateral inguinal hernioplasty.
3. That the surgery is performed in the Ambulatory Surgery Unit (UCA).

Exclusion Criteria:

1. Recurrent hernia.
2. allergies, ongoing infections, diabetes.
3. Background of rejection of prosthetic material (mesh).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
pain postoperative | 3 month
  It will be used a 10cm ruler which will allows the patients indicates how much pain they are feeling at the moment, where 0 is no pain at all and 10 is the maximum imaginable pain.

SECONDARY OUTCOMES:
take analgesic | 1 month
  Medication journal completed by patient

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian SR Roche, doctor, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Peron 4190, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Yes